CLINICAL TRIAL: NCT00048347
Title: An Open-Label, Pilot Study of Type I Interferon (AVONEX) Treatment of Ulcerative Colitis
Brief Title: Interferon-beta1a (AVONEX) Treatment of Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Peter Mannon, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030019; 03-I-0019 (Registry Identifier: NCT00048347)
Record Dates: First submitted 2002-10-29; First posted 2002-10-30 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-08

CONDITIONS: Ulcerative Colitis
Keywords: Lymphocyte; Monocyte; Inflammation; Th2; Colonoscopy; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammation | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avonex (Experimental): Interferon-beta1a (Avonex) 30 µg IM every week for 12 weeks
  Interventions: Drug: AVONEX

INTERVENTIONS:
Drug: AVONEX — 30µg IM every week for 12 weeks

SUMMARY:
This study will evaluate the safety and effectiveness of the drug interferon-beta1a (AVONEX) in treating ulcerative colitis and examine the drug's effect on the immune system. People with ulcerative colitis have increased amounts of inflammatory chemicals (cytokines) made by immune cells in the lining of the colon. Studies have shown that interferon-beta may block the activity of these cytokines. Interferon-beta1a (AVONEX) is currently FDA-approved to treat multiple sclerosis, a disease involving inflammation of the brain and spinal cord.

Patients 18 years of age and older who have had ulcerative colitis for at least 4 months may be eligible for this study. Candidates will be screened with a review of their medical records, a medical history and physical examination, electrocardiogram (EKG), blood, urine, and stool tests, and a pregnancy test for women of childbearing potential. A colonoscopy will also be done to determine disease activity and extent. This test uses a lighted tube to examine the amount of inflammation in the colon and take tissue samples (biopsies) for testing. Before the test, the patient is given a medicine to allay anxiety and the discomfort of inserting the endoscope into the rectum. This flexible tube allows the doctor to see the intestinal mucosa and project an image of the inner lining of the intestine onto a TV monitor. At various places in the intestine, small pieces of tissue are plucked out by a special device at the tip of the endoscope. The procedure generally lasts 30 minutes to 1 hour.

Participants will come to the NIH Clinical Center once a week for 4 weeks to receive an injection of interferon-beta, fill out questionnaires, and have a symptoms check, physical examination, and blood tests. Patients whose colitis has not worsened at the end of the 4 weeks and who have not had significant drug side effects will continue to receive weekly injections for an additional 8 weeks. Some patients may receive some of the last eight injections outside of NIH, but all patients will visit the Clinical Center visits every 3 to 4 weeks for a physical exam, symptoms check and blood tests.

After the 12 injections are completed, patients will have another colonoscopy to evaluate the response to treatment and will return to the Clinical Center every 6 weeks for a total of four visits, for a physical examination, symptoms check and blood tests.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the immunologic and clinical response to type I interferon administered to patients with ulcerative colitis. Ulcerative colitis (UC) is a chronic, relapsing inflammation of the colonic mucosa with major symptoms of diarrhea, hematochezia, abdominal pain, and an accompanying increase in colorectal carcinoma risk. Novel approaches to therapy of UC are required because the burden of disease is great (about 500,000 prevalent cases in the United States), standard medical therapy is limited in effectiveness and toxicity, and surgical therapy, albeit curative, results in permanent ostomies or complication-prone alternatives.

The rationale for this study is based on the observation that the mucosal inflammation in UC may be mediated by Th2 cytokines such as IL-4 or cytokines induced along with IL-4. Type I interferons can block IL-4 receptor signaling by up-regulating cytosolic inhibitory proteins (suppressor of cytokines signaling or SOCS proteins). Furthermore, two small studies of type I interferon effects on UC show benefit as opposed to many more studies in Crohn's disease, a classic Th1 inflammatory disease, which have shown no benefit from type I interferons. We hypothesize that type I interferons could be used to inhibit the pro-inflammatory signals of Th2 cytokines in UC.

This study will measure the immunologic and clinical effect of twelve weeks of treatment with a type I interferon administered to patients with active UC. The primary outcomes include documenting changes in immune parameters by measuring peripheral and lamina propria mononuclear cell cytokine release, expression levels of SOCS proteins in mononuclear cells, and changes in clinical parameters using the Short Clinical Colitis Activity Index and endoscopic and histologic scores. Secondary endpoints include the rate and severity of adverse events. Our short-term goal is to correlate changes in immune and biochemical parameters that accompany or predict clinical responses. The long-term goal of this study is to establish type I interferons as an effective alternative or adjunctive therapy with a low risk profile for the treatment of ulcerative colitis.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 years old or greater.
  2. Diagnosis of ulcerative colitis for at least 4 months based on endoscopic appearance or radiographic distribution of disease and corroborated with histopathology (especially the absence of granulomata).
  3. Presence of current active disease as defined by a Simple Clinical Colitis Activity Index of greater than or equal to 5 (for either of the two measurements done during the Screening Phase and that the second measurement is within 50 percent of the value of the first) who may or may not have the presence of one of the following: current corticosteroid- dependence for disease treatment, disease refractory to corticosteroids, or history of intolerance to treatment with corticosteroids (for criterion of co-administered corticosteroid dose see below).

     Corticosteroid-dependence is defined as relapse of ulcerative colitis within 60 days of completing a course of corticosteroid treatment, or during corticosteroid tapering at doses greater than or equal to 10 mg prednisone/day (or equivalent), or within three months following corticosteroid tapering while receiving a steroid dose of greater than or equal to 10 mg prednisone/day (or equivalent).
  4. If currently receiving medication for ulcerative colitis, patients may be on a stable regimen of one or a combination of the following drug doses and durations:

Corticosteroids (less than or equal to 25 mg Prednisone/d or Prednisone equivalent) is greater than or equal to 4 weeks;

5-ASA/Sulfasalazine is greater than or equal to 4 weeks;

Azathioprine/6-MP/thioguanine is greater than or equal to 12 weeks. (Note: Patients receiving azathioprine/6-MP/thioguanine must have been on a stable dose of this medication for greater than or equal to 8 weeks before randomization);

Probiotics (live bacterial dietary supplements) greater than or equal to 4 weeks;

Prebiotics (dietary supplements to produce biologically active substances) greater than or equal to 4 weeks.

5. Use of barrier or hormonal methods of birth control for female subjects who are not surgically sterile or postmenopausal.

6. Negative serum beta-hCG for women of child-bearing potential (women who are not surgically sterile or postmenopausal) to exclude early unnoticed pregnancy.

7. Negative results on stool examination for culture of enteric pathogens (Salmonella, Shigella, Yersinia, Campylobacter, Vibrio, E. coli O157/H7), Clostridium difficile toxin assay, enteric parasites and their ova (including Giardia and Cryptosporidia).

8. Thyroid function test and TSH level within establish normal range set by the Clinical Center.

EXCLUSION CRITERIA:

1. Inability to meet any of the above inclusion criteria.
2. Use of any of the following medications within the specified time period prior to the first dose of interferon-beta or at any time during the study:

   Non-steroidal anti-inflammatory agents (including COX-2 inhibitors), - 1 week

   Corticosteroids (greater than 25 mg Prednisone/d or Prednisone equivalent), Methotrexate, Cyclosporin, Tacrolimus, Thalidomide, or Mycophenolate mofetil - 4 weeks

   Monoclonal antibodies to TNF alpha or any Other Biologic (cytokine, anti-cytokine, or integrin-based therapy, for instance) - 4 months

   Any experimental agent - 1 month

   Concomitant use of any of the following drugs: isoniazid, iproniazid, dantrolene, ticrynafen (tienilic acid), ibufenac, bromfenac, benoxaprofen, zileutan, nicotinic acid, trovafloxacin, perhexiline, dilevavol, labetalol, pemoline, felbamate, tolcapone, diclofenac, AIDS drugs (HIV+ subjects are excluded anyway), and troglitozone.
3. History of colectomy, partial colectomy, current ostomy, or pouchitis.
4. Presence of significant electrocardiogram abnormalities including QT(c) greater than or equal to 0.48 sec, Mobitz type II second degree or third degree atrioventricular block, left bundle branch block or right bundle branch block accompanied by any fascicular block, changes consistent with acute ischemia or pericarditis.
5. Presence of a diagnosis of Crohn's disease, indeterminate colitis, microscopic colitis, ischemic colitis, or colitis attributable to infection. This determination may require use of clinical, endoscopic, and histologic data.
6. Presence of Cushing's syndrome.
7. Presence of current active bowel obstruction, intestinal perforation, significant GI hemorrhage, known presence of high grade stricture, history of toxic megacolon, history of colonic epithelium high-grade dysplasia or a dysplasia-associated lesion or mass that does not resemble an adenoma (that is a mass lesion, stricture, or broad-based tumor).
8. Anticipation that surgery may be required to treat the ulcerative colitis within 3 months of study entry.
9. HIV positivity or signs and symptoms consistent with HIV infection.
10. Acute systemic or intestinal infection requiring antibiotics.
11. Active hepatitis B or C.
12. Decompensated liver disease (Childs-Pugh class B or C).
13. Hematocrit less than 30 percent

    Platelet count 120,000 less than or greater than 850,000

    PT INR greater than 1.3 or PTT prolonged by greater than 3 seconds

    Serum creatinine or BUN greater than 1.5 times the upper limit of normal (ULN)

    ALT (SGPT) or AST (SGOT) greater than 2 times the ULN

    Total bilirubin greater than 1.25 times the ULN

    Alkaline phosphatase greater than 1.5 times the ULN.
14. Pregnancy or nursing (for women).
15. History of cancer (other than resected cutaneous basal or squamous cell carcinoma and in situ cervical cancer) with less than 5 years' documentation of a disease-free state.
16. History of a myocardial infarction within the last 12 months.
17. Any other condition that in the investigator's opinion places the patient at undue risk by participating in the study. This includes but is not limited to: psoriasis, thyroid disease, myasthenia gravis, lupus erythematosus, rheumatoid arthritis, Raynaud's disease, autoimmune hepatitis, C1 esterase deficiency or any deficiency of the complement system, and plasma cell dyscrasias.
18. History of anaphylactic reaction or hypersensitivity to natural or recombinant interferon-beta, human albumin, or proteins derived from CHO cells/formulation.
19. History of depression with psychotic features, or requiring ECT or hospitalization, or accompanied by suicidal ideation, gestures, or attempts.
20. History of seizure, except for isolated febrile seizure of childhood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-10; Primary Completion 2008-06 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Mannon, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Duchmann R, May E, Heike M, Knolle P, Neurath M, Meyer zum Buschenfelde KH. T cell specificity and cross reactivity towards enterobacteria, bacteroides, bifidobacterium, and antigens from resident intestinal flora in humans. Gut. 1999 Jun;44(6):812-8. doi: 10.1136/gut.44.6.812. PMID 10323882

RESULTS

PARTICIPANT FLOW:
Groups:
- Avonex: 30 µg IM every week for 12 weeks
Period: Overall Study
Arm/Group | Avonex
Started | 18
Completed | 16
Not Completed | 2
Not completed — Screen failure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Avonex
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 16
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 39.4 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With at Least a 3 Point Drop in the Short Clinical Colitis Score (SCCAI)
Description: The primary endpoint is the percent of patients with a clinical response as defined by a drop in the Short Clinical Colitis Score (SCCAI) of at least 3 points from Week 0 to Week 12. Short Clinical Colitis Score (SCCAI): Bowel frequency(day0-3,night0-2),urgency(0-3),rectal bleeding(0-3),well being(0-4),extracolonic features(0-4), total score 0(best)-19(worst).
Time Frame: Baseline, Week 12
Measure: Number; unit: Percent of participants
Arm/Group | Avonex
Number analyzed (Participants) | 18
Percent of participants | 63

ADVERSE EVENTS:
Arm/Group | Avonex
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 12/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avonex (N=16)
fever (Gastrointestinal disorders) | 10 (10) — Patients reported fever (63%) and mild flu-like symptoms (myalgias in 31%) after injections, but these were transient (usually resolving 4-5 hours after the injection) and responded well to treatment with acetominophen.
eosinophilia (Blood and lymphatic system disorders) | 1 (1)
paresthesias (Nervous system disorders) | 1 (1)
epistaxis (Blood and lymphatic system disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
pilonidal cyst (Infections and infestations) | 1 (1)
palmar xeroderma (Skin and subcutaneous tissue disorders) | 1 (1)
C. difficile colitis (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
While this study was designed as a proof-of-concept pilot trial to correlate changes in IL-13 and other cytokines with clinical response, efficacy was measured. The efficacy estimate is limited by the open-label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes